CLINICAL TRIAL: NCT00510042
Title: National Study of Moderate and Severe Von Willebrand Disease in the Netherlands
Acronym: WiN
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Foundation Haemophilia (Unknown); CSL Behring (Industry)
Responsible Party: F.W.G. Leebeek, MD PhD, Erasmus University Medical Center
Other Study IDs: MEC-2007-063
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Von Willebrand Disease
Keywords: von Willebrand disease; von Willebrand factor; national study; bleeding disorder; quality of life
MeSH Terms: conditions — von Willebrand Diseases; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma, DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to assess the clinical presentation, the treatment and the complications of the disease and treatment in moderate and severe von Willebrand disease. Another goal is to investigate the influence of von Willebrand disease on quality of life.

DETAILED DESCRIPTION:
The incidence of von Willebrand disease in the Netherlands is unknown, but the occurrence of all types of von Willebrand disease together is estimated at 1:100-1:200 individuals. Most patients have mild von Willebrand disease, mostly type 1. For the more severe forms of von Willebrand disease the incidence in unclear, but the expectation is, that there are at least 500-1500 patients. In the Netherlands, an unique situation exists for the treatment of patients with hemophilia and related coagulation disorders. In 2000 a hemophilia management policy was set up by the Ministry of Health, which stated that the care for these patients should be concentrated in 13 Hemophilia Treatment Centers (HTC). The representatives of the attending centers, the hemophilia specialists, are organized in the NVHB, the Dutch society of Hemophilia treaters. In the hemophilia management policy is stated that all patients with a coagulation disorder dependent of replacement products must be treated in a HTC or under responsibility of a HTC. These patients are seen in a HTC at least once a year.

Because all moderate and severe von Willebrand patients in the Netherlands are known in HTC, it is possible to register and study this population. This is imperative to the research of von Willebrand disease. Because the moderate and severe forms of von Willebrand disease are rare, it is impossible for an individual center to perform research of moderate severe and severe von Willebrand disease. Therefore a national approach is necessary.

For optimal care of patients with the moderate and severe form of von Willebrand disease a better understanding of symptoms, diagnostics, treatment and complications of treatment is necessary. The present study aims to register and investigate all patients in the Netherlands with moderate and severe von Willebrand disease to gain understanding of the clinical presentation, the treatment and the complications of treatment in moderate and severe von Willebrand disease. Another goal is to investigate the influence of von Willebrand disease on quality of life.

To answer these questions a questionnaire is developed, which will be sent to the study population. In addition, blood will be drawn for von Willebrand factor measurement and plasma and DNA will be stored. The relationship between laboratory parameters, (including von Willebrand factor, FVIII and prothrombotic coagulation disorders) and the clinical phenotype in patients with moderate and severe von Willebrand disease will be studied. We will assess the effect of the laboratory parameters on both the severity of bleeding tendency, and the possible protecting effect on the risk of arterial thrombosis. In the future mutation analysis of the VWF gene will be performed in patients with moderate and severe von Willebrand disease in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

1. haemorrhagic symptoms or a family history of von Willebrand disease
2. vWF antigen ≤ 30%, lowest measurement counts and/or vWF activity (vWF:RCo of vWF:CB) ≤ 30%, lowest measurement counts and/or FVIII:C ≤ 40 %, lowest measurement counts
3. being known in a hemophilia treatment center or if only the diagnose is made in a hemophilia treatment center this must be done after 1987

Exclusion Criteria:

1. Hemophilia A
2. Carriership of hemophilia A
3. No informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate and devere von Willebrand disease, known in a hemophilia treatment center
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2007-07; Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva M de Wee, MD, Study Director — Erasmus Medical Center; Frank WG Leebeek, MD, PhD, Principal Investigator — Erasmus Medical Center; Karin Fijn van Draat, MD, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Jeroen CJ Eikenboom, MD, PhD, Study Chair — Leiden University Medical Center; Arja de Goede-Bolder, MD, Study Chair — Erasmus Medical Center; Eveline P Mauser-Bunschoten, MD, PhD, Study Chair — Van Creveldkliniek, University Medical Center Utrecht; Karina Meijer, MD, PhD, Study Chair — University Medical Center Goningen; Britta Laros-van Gorkom, MD, PhD, Study Chair — University Medical Center St. Radboud Nijmegen; Johanna G van der Bom, PhD, Study Chair — Leiden University Medical Center; Manon A Degenaar-Dujardin, BA, Study Chair — Organization for Hemophilia Patients
Locations (12):
- Netherlands (12):
  - Academic Medical Center Amsterdam, Amsterdam
  - VU University Medical Center, Amsterdam
  - Amphia Hospital, Breda
  - Maxima Medical Center, Eindhoven
  - University Medical Center Groningen, Groningen
  - Kennemer Hospital, Haarlem
  - Leiden University Medical Center, Leiden
  - Academic Hospital Maastricht, Maastricht
  - University Medical Center St. Radboud, Nijmegen
  - Erasmus University Medical Center, Rotterdam
  - Haga Hospital, The Hague
  - University Medical Center Utrecht Van Creveldkliniek, Utrecht

REFERENCES:
- [Background] Mannucci PM. Treatment of von Willebrand's Disease. N Engl J Med. 2004 Aug 12;351(7):683-94. doi: 10.1056/NEJMra040403. No abstract available. PMID 15306670
- [Background] Sadler JE, Mannucci PM, Berntorp E, Bochkov N, Boulyjenkov V, Ginsburg D, Meyer D, Peake I, Rodeghiero F, Srivastava A. Impact, diagnosis and treatment of von Willebrand disease. Thromb Haemost. 2000 Aug;84(2):160-74. No abstract available. PMID 10959685
- [Background] Sadler JE. A revised classification of von Willebrand disease. For the Subcommittee on von Willebrand Factor of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Thromb Haemost. 1994 Apr;71(4):520-5. PMID 8052974
- [Background] Tosetto A, Rodeghiero F, Castaman G, Goodeve A, Federici AB, Batlle J, Meyer D, Fressinaud E, Mazurier C, Goudemand J, Eikenboom J, Schneppenheim R, Budde U, Ingerslev J, Vorlova Z, Habart D, Holmberg L, Lethagen S, Pasi J, Hill F, Peake I. A quantitative analysis of bleeding symptoms in type 1 von Willebrand disease: results from a multicenter European study (MCMDM-1 VWD). J Thromb Haemost. 2006 Apr;4(4):766-73. doi: 10.1111/j.1538-7836.2006.01847.x. PMID 16634745
- [Background] Federici AB. Clinical diagnosis of von Willebrand disease. Haemophilia. 2004 Oct;10 Suppl 4:169-76. doi: 10.1111/j.1365-2516.2004.00991.x. PMID 15479393